CLINICAL TRIAL: NCT01155570
Title: Special Investigation (All Cases Investigation in Patients With Psoriasis Vulgaris and Psoriatic Arthritis)
Brief Title: Special Investigation in Patients With Psoriasis Vulgaris and Psoriatic Arthritis (All Patients Investigation)
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-077
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Results first posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Humira: Humira 40 mg (marketed product) every other week (eow) for subcutaneous injection after initial dosage of 80 mg.

SUMMARY:
The survey will be conducted with regard to the following aspects of treatment with Humira (adalimumab) in patients with psoriasis vulgaris and psoriatic arthritis receiving this drug:

* unknown adverse drug reactions, especially clinically significant adverse reactions
* incidence and conditions of occurrence of adverse reactions in the clinical setting
* factors that may affect the safety and effectiveness of Humira.

DETAILED DESCRIPTION:
This study was non-interventional, open-labeled, all-cases, central registration method, post marketing observational study in which Humira was prescribed for patients with psoriasis vulgaris and/or psoriatic arthritis in routine medical practice.

When investigators prescribed Humira to an eligible patient who provided informed consent, they filled out a registration form and send it to the registration center via postal mail. At the end of the 24-week observation period, an investigator filled out a case report form for each patient to describe the findings during the study period, and provided the completed form to medical representatives. Even if Humira treatment was for any reason discontinued, the investigators followed each such participant for 24 weeks after the first administration of Humira, and filled out a case report form for the participant at the end of the 24-week period.

Some participants entered this study from study NCT00647400 (M04-702), a Phase III extension study of Humira (adalimumab) in Japan.

ELIGIBILITY:
Inclusion Criteria:

All patients who receive Humira for the treatment of psoriasis vulgaris or psoriatic arthritis not responding to conventional treatment will be evaluated. Eligible patients should be

* those not responding to at least one type of conventional systemic treatment (including ultraviolet therapy) who have skin lesions involving 10% of body surface area or
* patients with intractable eruptions of joint signs/symptoms.

Exclusion Criteria:

Contraindications according to the Package Insert include patients who have any of the following:

* serious infections
* tuberculosis
* a history of hypersensitivity to any ingredient of Humira
* demyelinating disease or a history of demyelinating disease
* congestive cardiac failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who receive Humira for the treatment of psoriasis vulgaris or psoriatic arthritis
Sampling Method: Non-Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Yamaguchi, MD, Study Director — AbbVie
Locations (634):
- Japan (634):
  - Site Reference ID/Investigator# 41606, Aichi
  - Site Reference ID/Investigator# 41769, Aichi
  - Site Reference ID/Investigator# 41810, Aichi
  - Site Reference ID/Investigator# 56131, Aichi
  - Site Reference ID/Investigator# 56251, Aichi
  - Site Reference ID/Investigator# 56252, Aichi
  - Site Reference ID/Investigator# 56254, Aichi
  - Site Reference ID/Investigator# 56340, Aichi
  - Site Reference ID/Investigator# 60016, Aichi
  - Site Reference ID/Investigator# 67150, Aichi
  - Site Reference ID/Investigator# 68627, Aichi
  - Site Reference ID/Investigator# 41327, Aizu-Wakamatsu
  - Site Reference ID/Investigator# 41820, Akita
  - Site Reference ID/Investigator# 41823, Akita
  - Site Reference ID/Investigator# 41684, Amagasaki
  - Site Reference ID/Investigator# 41851, Amagasaki
  - Site Reference ID/Investigator# 41305, Anjo
  - Site Reference ID/Investigator# 41822, Aomori
  - Site Reference ID/Investigator# 60012, Aomori
  - Site Reference ID/Investigator# 64811, Aomori
  - Site Reference ID/Investigator# 41800, Asahikawa
  - Site Reference ID/Investigator# 80887, Ashikaga
  - Site Reference ID/Investigator# 80879, Ayabe
  - Site Reference ID/Investigator# 41207, Bunkyo-ku, Tokyo
  - Site Reference ID/Investigator# 41247, Chiba
  - Site Reference ID/Investigator# 41258, Chiba
  - Site Reference ID/Investigator# 41260, Chiba
  - Site Reference ID/Investigator# 41263, Chiba
  - Site Reference ID/Investigator# 41485, Chiba
  - Site Reference ID/Investigator# 41821, Chiba
  - Site Reference ID/Investigator# 41927, Chiba
  - Site Reference ID/Investigator# 56127, Chiba
  - Site Reference ID/Investigator# 56224, Chiba
  - Site Reference ID/Investigator# 59995, Chiba
  - Site Reference ID/Investigator# 41893, Chūō
  - Site Reference ID/Investigator# 41721, Ehime
  - Site Reference ID/Investigator# 41724, Ehime
  - Site Reference ID/Investigator# 41727, Ehime
  - Site Reference ID/Investigator# 80873, Fujieda
  - Site Reference ID/Investigator# 41287, Fujisawa
  - Site Reference ID/Investigator# 41550, Fukui
  - Site Reference ID/Investigator# 41693, Fukui
  - Site Reference ID/Investigator# 41694, Fukui
  - Site Reference ID/Investigator# 41697, Fukui
  - Site Reference ID/Investigator# 41746, Fukui
  - Site Reference ID/Investigator# 41805, Fukui
  - Site Reference ID/Investigator# 41326, Fukuoka
  - Site Reference ID/Investigator# 41476, Fukuoka
  - Site Reference ID/Investigator# 41604, Fukuoka
  - Site Reference ID/Investigator# 41607, Fukuoka
  - Site Reference ID/Investigator# 41731, Fukuoka
  - Site Reference ID/Investigator# 41734, Fukuoka
  - Site Reference ID/Investigator# 41747, Fukuoka
  - Site Reference ID/Investigator# 41796, Fukuoka
  - Site Reference ID/Investigator# 41812, Fukuoka
  - Site Reference ID/Investigator# 56349, Fukuoka
  - Site Reference ID/Investigator# 56350, Fukuoka
  - Site Reference ID/Investigator# 59987, Fukuoka
  - Site Reference ID/Investigator# 59991, Fukuoka
  - Site Reference ID/Investigator# 41745, Fukushima
  - Site Reference ID/Investigator# 41757, Fukushima
  - Site Reference ID/Investigator# 41758, Fukushima
  - Site Reference ID/Investigator# 41818, Fukushima
  - Site Reference ID/Investigator# 41824, Fukushima
  - Site Reference ID/Investigator# 41825, Fukushima
  - Site Reference ID/Investigator# 56095, Fukushima
  - Site Reference ID/Investigator# 56242, Fukushima
  - Site Reference ID/Investigator# 56330, Fukushima
  - Site Reference ID/Investigator# 41301, Gifu
  - Site Reference ID/Investigator# 41302, Gifu
  - Site Reference ID/Investigator# 41306, Gifu
  - Site Reference ID/Investigator# 41309, Gifu
  - Site Reference ID/Investigator# 41322, Gifu
  - Site Reference ID/Investigator# 41774, Gifu
  - Site Reference ID/Investigator# 56103, Gifu
  - Site Reference ID/Investigator# 59989, Gifu
  - Site Reference ID/Investigator# 41830, Gunma
  - Site Reference ID/Investigator# 56122, Gunma
  - Site Reference ID/Investigator# 56123, Gunma
  - Site Reference ID/Investigator# 56207, Gunma
  - Site Reference ID/Investigator# 59986, Gunma
  - Site Reference ID/Investigator# 59997, Gunma
  - Site Reference ID/Investigator# 41828, Hakodate
  - Site Reference ID/Investigator# 41303, Hamamatsu
  - Site Reference ID/Investigator# 41304, Hamamatsu
  - Site Reference ID/Investigator# 59992, Hamamatsu
  - Site Reference ID/Investigator# 80895, Hamamatsu
  - Site Reference ID/Investigator# 56135, Hannan
  - Site Reference ID/Investigator# 56198, Higashihiroshima
  - Site Reference ID/Investigator# 41748, Himeji
  - Site Reference ID/Investigator# 41917, Himeji
  - Site Reference ID/Investigator# 41668, Hirakata
  - Site Reference ID/Investigator# 41915, Hirosaki
  - Site Reference ID/Investigator# 41712, Hiroshima
  - Site Reference ID/Investigator# 41713, Hiroshima
  - Site Reference ID/Investigator# 41714, Hiroshima
  - Site Reference ID/Investigator# 41715, Hiroshima
  - Site Reference ID/Investigator# 41716, Hiroshima
  - Site Reference ID/Investigator# 41717, Hiroshima
  - Site Reference ID/Investigator# 41753, Hiroshima
  - Site Reference ID/Investigator# 41773, Hiroshima
  - Site Reference ID/Investigator# 41833, Hiroshima
  - Site Reference ID/Investigator# 41835, Hiroshima
  - Site Reference ID/Investigator# 56196, Hiroshima
  - Site Reference ID/Investigator# 56197, Hiroshima
  - Site Reference ID/Investigator# 56346, Hiroshima
  - Site Reference ID/Investigator# 56347, Hiroshima
  - Site Reference ID/Investigator# 59988, Hiroshima
  - Site Reference ID/Investigator# 59999, Hiroshima
  - Site Reference ID/Investigator# 60013, Hiroshima
  - Site Reference ID/Investigator# 60017, Hiroshima
  - Site Reference ID/Investigator# 60018, Hiroshima
  - Site Reference ID/Investigator# 41827, Hokkaido
  - Site Reference ID/Investigator# 41829, Hokkaido
  - Site Reference ID/Investigator# 41832, Hokkaido
  - Site Reference ID/Investigator# 41837, Hokkaido
  - Site Reference ID/Investigator# 41838, Hokkaido
  - Site Reference ID/Investigator# 41842, Hokkaido
  - Site Reference ID/Investigator# 41844, Hokkaido
  - Site Reference ID/Investigator# 41847, Hokkaido
  - Site Reference ID/Investigator# 41852, Hokkaido
  - Site Reference ID/Investigator# 41929, Hokkaido
  - Site Reference ID/Investigator# 56109, Hokkaido
  - Site Reference ID/Investigator# 56206, Hokkaido
  - Site Reference ID/Investigator# 56327, Hokkaido
  - Site Reference ID/Investigator# 60014, Hokkaido
  - Site Reference ID/Investigator# 64802, Hokkaido
  - Site Reference ID/Investigator# 64813, Hokkaido
  - Site Reference ID/Investigator# 67144, Hokkaido
  - Site Reference ID/Investigator# 71456, Hokkaido
  - Site Reference ID/Investigator# 41481, Hyōgo
  - Site Reference ID/Investigator# 41683, Hyōgo
  - Site Reference ID/Investigator# 41687, Hyōgo
  - Site Reference ID/Investigator# 41691, Hyōgo
  - Site Reference ID/Investigator# 41750, Hyōgo
  - Site Reference ID/Investigator# 41771, Hyōgo
  - Site Reference ID/Investigator# 41846, Hyōgo
  - Site Reference ID/Investigator# 56142, Hyōgo
  - Site Reference ID/Investigator# 56143, Hyōgo
  - Site Reference ID/Investigator# 56144, Hyōgo
  - Site Reference ID/Investigator# 56146, Hyōgo
  - Site Reference ID/Investigator# 56342, Hyōgo
  - Site Reference ID/Investigator# 56343, Hyōgo
  - Site Reference ID/Investigator# 60015, Hyōgo
  - Site Reference ID/Investigator# 67149, Hyōgo
  - Site Reference ID/Investigator# 41848, Ibaraki
  - Site Reference ID/Investigator# 41849, Ibaraki
  - Site Reference ID/Investigator# 41858, Ibaraki
  - Site Reference ID/Investigator# 41908, Ichikawa
  - Site Reference ID/Investigator# 41293, Ichinomiya
  - Site Reference ID/Investigator# 56229, Ichinomiya
  - Site Reference ID/Investigator# 56333, Ichinomiya
  - Site Reference ID/Investigator# 41696, Iijima
  - Site Reference ID/Investigator# 56137, Ikoma
  - Site Reference ID/Investigator# 56226, Inabe
  - Site Reference ID/Investigator# 56120, Inashiki
  - Site Reference ID/Investigator# 80893, Inzai
  - Site Reference ID/Investigator# 41740, Isahaya
  - Site Reference ID/Investigator# 56230, Isesaki
  - Site Reference ID/Investigator# 41330, Ishikawa
  - Site Reference ID/Investigator# 41543, Ishikawa
  - Site Reference ID/Investigator# 41695, Ishikawa
  - Site Reference ID/Investigator# 41920, Ishikawa
  - Site Reference ID/Investigator# 41889, Iwafune
  - Site Reference ID/Investigator# 56348, Iwakuni
  - Site Reference ID/Investigator# 80916, Iwakuni
  - Site Reference ID/Investigator# 41704, Izumo
  - Site Reference ID/Investigator# 41719, Izumo
  - Site Reference ID/Investigator# 56195, Izumo
  - Site Reference ID/Investigator# 41294, Izunokuni
  - Site Reference ID/Investigator# 41299, Izunokuni
  - Site Reference ID/Investigator# 41300, Izunokuni
  - Site Reference ID/Investigator# 60006, Jōetsu
  - Site Reference ID/Investigator# 41720, Kagawa
  - Site Reference ID/Investigator# 41725, Kagawa
  - Site Reference ID/Investigator# 56200, Kagawa
  - Site Reference ID/Investigator# 56201, Kagawa
  - Site Reference ID/Investigator# 41737, Kagoshima
  - Site Reference ID/Investigator# 67145, Kagoshima
  - Site Reference ID/Investigator# 41283, Kanagawa
  - Site Reference ID/Investigator# 41284, Kanagawa
  - Site Reference ID/Investigator# 41451, Kanagawa
  - Site Reference ID/Investigator# 41452, Kanagawa
  - Site Reference ID/Investigator# 41815, Kanagawa
  - Site Reference ID/Investigator# 41854, Kanagawa
  - Site Reference ID/Investigator# 41856, Kanagawa
  - Site Reference ID/Investigator# 41862, Kanagawa
  - Site Reference ID/Investigator# 56098, Kanagawa
  - Site Reference ID/Investigator# 56250, Kanagawa
  - Site Reference ID/Investigator# 60011, Kanagawa
  - Site Reference ID/Investigator# 64805, Kanagawa
  - Site Reference ID/Investigator# 68629, Kanagawa
  - Site Reference ID/Investigator# 41699, Kanazawa
  - Site Reference ID/Investigator# 41762, Kariya
  - Site Reference ID/Investigator# 41461, Kashihara
  - Site Reference ID/Investigator# 41486, Kashiwa
  - Site Reference ID/Investigator# 41482, Kawagoe
  - Site Reference ID/Investigator# 41484, Kawagoe
  - Site Reference ID/Investigator# 41784, Kawagoe
  - Site Reference ID/Investigator# 41279, Kawasaki
  - Site Reference ID/Investigator# 41280, Kawasaki
  - Site Reference ID/Investigator# 41281, Kawasaki
  - Site Reference ID/Investigator# 41282, Kawasaki
  - Site Reference ID/Investigator# 71453, Kawasaki
  - Site Reference ID/Investigator# 80880, Kawasaki
  - Site Reference ID/Investigator# 41269, Kisarazu
  - Site Reference ID/Investigator# 41733, Kitakyushu
  - Site Reference ID/Investigator# 41735, Kitakyushu
  - Site Reference ID/Investigator# 68626, Kitakyushu
  - Site Reference ID/Investigator# 71454, Kitakyushu
  - Site Reference ID/Investigator# 80892, Kitakyushu
  - Site Reference ID/Investigator# 41471, Kobe
  - Site Reference ID/Investigator# 41472, Kobe
  - Site Reference ID/Investigator# 41544, Kobe
  - Site Reference ID/Investigator# 41686, Kobe
  - Site Reference ID/Investigator# 56090, Kobe
  - Site Reference ID/Investigator# 56145, Kobe
  - Site Reference ID/Investigator# 56264, Kobe
  - Site Reference ID/Investigator# 80874, Kobe
  - Site Reference ID/Investigator# 80883, Kobe
  - Site Reference ID/Investigator# 80914, Kobe
  - Site Reference ID/Investigator# 41480, Kochi
  - Site Reference ID/Investigator# 41548, Kochi
  - Site Reference ID/Investigator# 89493, Kofu
  - Site Reference ID/Investigator# 60003, Komaki
  - Site Reference ID/Investigator# 67153, Komoro
  - Site Reference ID/Investigator# 41262, Koshigaya
  - Site Reference ID/Investigator# 41817, Kōnan
  - Site Reference ID/Investigator# 41798, Kōriyama
  - Site Reference ID/Investigator# 41819, Kōriyama
  - Site Reference ID/Investigator# 64808, Kōtari
  - Site Reference ID/Investigator# 56263, Kudamatsu
  - Site Reference ID/Investigator# 56087, Kumamoto
  - Site Reference ID/Investigator# 56351, Kumamoto
  - Site Reference ID/Investigator# 41467, Kurashiki
  - Site Reference ID/Investigator# 41903, Kurashiki
  - Site Reference ID/Investigator# 41904, Kurashiki
  - Site Reference ID/Investigator# 41926, Kurashiki
  - Site Reference ID/Investigator# 60001, Kurashiki
  - Site Reference ID/Investigator# 41718, Kure
  - Site Reference ID/Investigator# 41689, Kurobe
  - Site Reference ID/Investigator# 41460, Kurume
  - Site Reference ID/Investigator# 56202, Kurume
  - Site Reference ID/Investigator# 41839, Kushiro
  - Site Reference ID/Investigator# 41454, Kyoto
  - Site Reference ID/Investigator# 41698, Kyoto
  - Site Reference ID/Investigator# 41700, Kyoto
  - Site Reference ID/Investigator# 41705, Kyoto
  - Site Reference ID/Investigator# 41768, Kyoto
  - Site Reference ID/Investigator# 41801, Kyoto
  - Site Reference ID/Investigator# 41806, Kyoto
  - Site Reference ID/Investigator# 41905, Kyoto
  - Site Reference ID/Investigator# 41921, Kyoto
  - Site Reference ID/Investigator# 56193, Kyoto
  - Site Reference ID/Investigator# 56194, Kyoto
  - Site Reference ID/Investigator# 56259, Kyoto
  - Site Reference ID/Investigator# 56344, Kyoto
  - Site Reference ID/Investigator# 60005, Kyoto
  - Site Reference ID/Investigator# 64807, Kyoto
  - Site Reference ID/Investigator# 41831, Maebashi
  - Site Reference ID/Investigator# 41834, Maebashi
  - Site Reference ID/Investigator# 56121, Maebashi
  - Site Reference ID/Investigator# 67263, Maebashi
  - Site Reference ID/Investigator# 59994, Maizuru
  - Site Reference ID/Investigator# 41900, Matsumoto
  - Site Reference ID/Investigator# 41901, Matsumoto
  - Site Reference ID/Investigator# 41324, Matsuyama
  - Site Reference ID/Investigator# 41723, Matsuyama
  - Site Reference ID/Investigator# 41902, Matsuyama
  - Site Reference ID/Investigator# 41308, Mie
  - Site Reference ID/Investigator# 41749, Mie
  - Site Reference ID/Investigator# 56208, Mie
  - Site Reference ID/Investigator# 56255, Mie
  - Site Reference ID/Investigator# 59996, Mie
  - Site Reference ID/Investigator# 41608, Minato
  - Site Reference ID/Investigator# 41794, Minato
  - Site Reference ID/Investigator# 41760, Mito
  - Site Reference ID/Investigator# 41855, Miyagi
  - Site Reference ID/Investigator# 41859, Miyagi
  - Site Reference ID/Investigator# 41861, Miyagi
  - Site Reference ID/Investigator# 41865, Miyagi
  - Site Reference ID/Investigator# 41871, Miyagi
  - Site Reference ID/Investigator# 56111, Miyagi
  - Site Reference ID/Investigator# 56112, Miyagi
  - Site Reference ID/Investigator# 56329, Miyagi
  - Site Reference ID/Investigator# 41475, Miyazaki
  - Site Reference ID/Investigator# 41790, Miyazaki
  - Site Reference ID/Investigator# 41791, Miyazaki
  - Site Reference ID/Investigator# 41919, Miyazaki
  - Site Reference ID/Investigator# 60021, Miyazaki
  - Site Reference ID/Investigator# 41458, Morioka
  - Site Reference ID/Investigator# 41462, Nagakute
  - Site Reference ID/Investigator# 41545, Nagakute
  - Site Reference ID/Investigator# 41797, Nagano
  - Site Reference ID/Investigator# 41863, Nagano
  - Site Reference ID/Investigator# 41866, Nagano
  - Site Reference ID/Investigator# 41870, Nagano
  - Site Reference ID/Investigator# 56124, Nagano
  - Site Reference ID/Investigator# 41464, Nagasaki
  - Site Reference ID/Investigator# 41728, Nagasaki
  - Site Reference ID/Investigator# 41730, Nagasaki
  - Site Reference ID/Investigator# 41736, Nagasaki
  - Site Reference ID/Investigator# 41756, Nagasaki
  - Site Reference ID/Investigator# 41789, Nagasaki
  - Site Reference ID/Investigator# 41864, Nagasaki
  - Site Reference ID/Investigator# 41877, Nagasaki
  - Site Reference ID/Investigator# 41289, Nagoya
  - Site Reference ID/Investigator# 41290, Nagoya
  - Site Reference ID/Investigator# 41549, Nagoya
  - Site Reference ID/Investigator# 41744, Nagoya
  - Site Reference ID/Investigator# 41802, Nagoya
  - Site Reference ID/Investigator# 41909, Nagoya
  - Site Reference ID/Investigator# 41910, Nagoya
  - Site Reference ID/Investigator# 56130, Nagoya
  - Site Reference ID/Investigator# 41804, Nanao
  - Site Reference ID/Investigator# 41478, Nankoku
  - Site Reference ID/Investigator# 41710, Nara
  - Site Reference ID/Investigator# 56091, Nara
  - Site Reference ID/Investigator# 56227, Nara
  - Site Reference ID/Investigator# 59985, Nara
  - Site Reference ID/Investigator# 80896, Nayori
  - Site Reference ID/Investigator# 67152, Nigata-honmachi
  - Site Reference ID/Investigator# 41793, Niigata
  - Site Reference ID/Investigator# 41873, Niigata
  - Site Reference ID/Investigator# 41879, Niigata
  - Site Reference ID/Investigator# 56326, Niigata
  - Site Reference ID/Investigator# 64812, Niigata
  - Site Reference ID/Investigator# 41741, Nishihara
  - Site Reference ID/Investigator# 41682, Nishinomiya
  - Site Reference ID/Investigator# 41690, Nishinomiya
  - Site Reference ID/Investigator# 80877, Nishio
  - Site Reference ID/Investigator# 67264, Nisshin
  - Site Reference ID/Investigator# 41914, Numakunai
  - Site Reference ID/Investigator# 59998, Numakunai
  - Site Reference ID/Investigator# 41841, Obihiro
  - Site Reference ID/Investigator# 41843, Obihiro
  - Site Reference ID/Investigator# 41857, Odawara
  - Site Reference ID/Investigator# 41701, Okayama
  - Site Reference ID/Investigator# 41702, Okayama
  - Site Reference ID/Investigator# 41703, Okayama
  - Site Reference ID/Investigator# 41709, Okayama
  - Site Reference ID/Investigator# 41918, Okayama
  - Site Reference ID/Investigator# 60019, Okayama
  - Site Reference ID/Investigator# 64809, Okayama
  - Site Reference ID/Investigator# 41310, Osaka
  - Site Reference ID/Investigator# 41455, Osaka
  - Site Reference ID/Investigator# 41456, Osaka
  - Site Reference ID/Investigator# 41466, Osaka
  - Site Reference ID/Investigator# 41477, Osaka
  - Site Reference ID/Investigator# 41662, Osaka
  - Site Reference ID/Investigator# 41663, Osaka
  - Site Reference ID/Investigator# 41664, Osaka
  - Site Reference ID/Investigator# 41667, Osaka
  - Site Reference ID/Investigator# 41669, Osaka
  - Site Reference ID/Investigator# 41670, Osaka
  - Site Reference ID/Investigator# 41671, Osaka
  - Site Reference ID/Investigator# 41672, Osaka
  - Site Reference ID/Investigator# 41673, Osaka
  - Site Reference ID/Investigator# 41674, Osaka
  - Site Reference ID/Investigator# 41675, Osaka
  - Site Reference ID/Investigator# 41676, Osaka
  - Site Reference ID/Investigator# 41678, Osaka
  - Site Reference ID/Investigator# 41679, Osaka
  - Site Reference ID/Investigator# 41680, Osaka
  - Site Reference ID/Investigator# 41743, Osaka
  - Site Reference ID/Investigator# 41786, Osaka
  - Site Reference ID/Investigator# 41799, Osaka
  - Site Reference ID/Investigator# 41809, Osaka
  - Site Reference ID/Investigator# 41811, Osaka
  - Site Reference ID/Investigator# 41874, Osaka
  - Site Reference ID/Investigator# 41875, Osaka
  - Site Reference ID/Investigator# 41878, Osaka
  - Site Reference ID/Investigator# 56088, Osaka
  - Site Reference ID/Investigator# 56134, Osaka
  - Site Reference ID/Investigator# 56205, Osaka
  - Site Reference ID/Investigator# 56256, Osaka
  - Site Reference ID/Investigator# 56257, Osaka
  - Site Reference ID/Investigator# 56325, Osaka
  - Site Reference ID/Investigator# 56341, Osaka
  - Site Reference ID/Investigator# 59990, Osaka
  - Site Reference ID/Investigator# 67143, Osaka
  - Site Reference ID/Investigator# 67148, Osaka
  - Site Reference ID/Investigator# 67151, Osaka
  - Site Reference ID/Investigator# 80878, Osaka
  - Site Reference ID/Investigator# 80882, Osaka
  - Site Reference ID/Investigator# 80915, Osaka
  - Site Reference ID/Investigator# 41766, Ōgaki
  - Site Reference ID/Investigator# 41906, Ōita
  - Site Reference ID/Investigator# 56203, Ōita
  - Site Reference ID/Investigator# 80876, Ōkawa
  - Site Reference ID/Investigator# 41840, Ōsaki
  - Site Reference ID/Investigator# 41867, Ōsaki
  - Site Reference ID/Investigator# 41869, Ōsaki
  - Site Reference ID/Investigator# 56113, Ōsaki
  - Site Reference ID/Investigator# 41708, Ōtsu
  - Site Reference ID/Investigator# 56345, Ōtsu
  - Site Reference ID/Investigator# 80875, Rifu
  - Site Reference ID/Investigator# 41729, Saga
  - Site Reference ID/Investigator# 41732, Saga
  - Site Reference ID/Investigator# 41876, Saga
  - Site Reference ID/Investigator# 41323, Sagamihara
  - Site Reference ID/Investigator# 41468, Sagamihara, Kanagawa
  - Site Reference ID/Investigator# 41256, Saitama
  - Site Reference ID/Investigator# 41257, Saitama
  - Site Reference ID/Investigator# 41261, Saitama
  - Site Reference ID/Investigator# 41264, Saitama
  - Site Reference ID/Investigator# 41265, Saitama
  - Site Reference ID/Investigator# 41266, Saitama
  - Site Reference ID/Investigator# 41267, Saitama
  - Site Reference ID/Investigator# 41270, Saitama
  - Site Reference ID/Investigator# 41271, Saitama
  - Site Reference ID/Investigator# 41272, Saitama
  - Site Reference ID/Investigator# 41274, Saitama
  - Site Reference ID/Investigator# 41278, Saitama
  - Site Reference ID/Investigator# 41329, Saitama
  - Site Reference ID/Investigator# 56094, Saitama
  - Site Reference ID/Investigator# 56099, Saitama
  - Site Reference ID/Investigator# 56100, Saitama
  - Site Reference ID/Investigator# 56249, Saitama
  - Site Reference ID/Investigator# 60009, Saitama
  - Site Reference ID/Investigator# 64803, Saitama
  - Site Reference ID/Investigator# 64804, Saitama
  - Site Reference ID/Investigator# 64810, Saitama
  - Site Reference ID/Investigator# 41603, Sakai
  - Site Reference ID/Investigator# 56136, Sakai
  - Site Reference ID/Investigator# 41868, Saku
  - Site Reference ID/Investigator# 41826, Sakura
  - Site Reference ID/Investigator# 41763, Sapporo
  - Site Reference ID/Investigator# 41850, Sapporo
  - Site Reference ID/Investigator# 41853, Sapporo
  - Site Reference ID/Investigator# 56105, Sapporo
  - Site Reference ID/Investigator# 56107, Sapporo
  - Site Reference ID/Investigator# 56108, Sapporo
  - Site Reference ID/Investigator# 56209, Sapporo
  - Site Reference ID/Investigator# 80884, Sapporo
  - Site Reference ID/Investigator# 41739, Sasebo
  - Site Reference ID/Investigator# 41755, Sasebo
  - Site Reference ID/Investigator# 41457, Sayama
  - Site Reference ID/Investigator# 41469, Sayama
  - Site Reference ID/Investigator# 41605, Sendai
  - Site Reference ID/Investigator# 41813, Sendai
  - Site Reference ID/Investigator# 41814, Sendai
  - Site Reference ID/Investigator# 41930, Sendai
  - Site Reference ID/Investigator# 80889, Sendai
  - Site Reference ID/Investigator# 41546, Seto
  - Site Reference ID/Investigator# 41553, Shiga
  - Site Reference ID/Investigator# 41707, Shiga
  - Site Reference ID/Investigator# 41754, Shiga
  - Site Reference ID/Investigator# 41922, Shiga
  - Site Reference ID/Investigator# 59993, Shiga
  - Site Reference ID/Investigator# 60007, Shimane
  - Site Reference ID/Investigator# 41884, Shimotsuke
  - Site Reference ID/Investigator# 41885, Shimotsuke
  - Site Reference ID/Investigator# 41292, Shizuoka
  - Site Reference ID/Investigator# 41295, Shizuoka
  - Site Reference ID/Investigator# 41296, Shizuoka
  - Site Reference ID/Investigator# 41298, Shizuoka
  - Site Reference ID/Investigator# 41328, Shizuoka
  - Site Reference ID/Investigator# 41479, Shizuoka
  - Site Reference ID/Investigator# 41772, Shizuoka
  - Site Reference ID/Investigator# 41808, Shizuoka
  - Site Reference ID/Investigator# 41872, Shizuoka
  - Site Reference ID/Investigator# 41880, Shizuoka
  - Site Reference ID/Investigator# 41881, Shizuoka
  - Site Reference ID/Investigator# 56101, Shizuoka
  - Site Reference ID/Investigator# 56132, Shizuoka
  - Site Reference ID/Investigator# 56133, Shizuoka
  - Site Reference ID/Investigator# 56253, Shizuoka
  - Site Reference ID/Investigator# 56339, Shizuoka
  - Site Reference ID/Investigator# 68628, Shizuoka
  - Site Reference ID/Investigator# 41928, Shūnan
  - Site Reference ID/Investigator# 80886, Sōka
  - Site Reference ID/Investigator# 41551, Takamatsu
  - Site Reference ID/Investigator# 41552, Takamatsu
  - Site Reference ID/Investigator# 41761, Takamatsu
  - Site Reference ID/Investigator# 41836, Takasaki
  - Site Reference ID/Investigator# 41665, Takatsuki
  - Site Reference ID/Investigator# 41666, Takatsuki
  - Site Reference ID/Investigator# 41767, Takatsuki
  - Site Reference ID/Investigator# 56138, Tanabe
  - Site Reference ID/Investigator# 41465, Tenri
  - Site Reference ID/Investigator# 41752, Tenri
  - Site Reference ID/Investigator# 41803, Tokushima
  - Site Reference ID/Investigator# 56222, Tokushima
  - Site Reference ID/Investigator# 67146, Tokushima
  - Site Reference ID/Investigator# 26162, Tokyo
  - Site Reference ID/Investigator# 41206, Tokyo
  - Site Reference ID/Investigator# 41208, Tokyo
  - Site Reference ID/Investigator# 41209, Tokyo
  - Site Reference ID/Investigator# 41210, Tokyo
  - Site Reference ID/Investigator# 41211, Tokyo
  - Site Reference ID/Investigator# 41212, Tokyo
  - Site Reference ID/Investigator# 41213, Tokyo
  - Site Reference ID/Investigator# 41214, Tokyo
  - Site Reference ID/Investigator# 41222, Tokyo
  - Site Reference ID/Investigator# 41223, Tokyo
  - Site Reference ID/Investigator# 41224, Tokyo
  - Site Reference ID/Investigator# 41225, Tokyo
  - Site Reference ID/Investigator# 41226, Tokyo
  - Site Reference ID/Investigator# 41227, Tokyo
  - Site Reference ID/Investigator# 41228, Tokyo
  - Site Reference ID/Investigator# 41229, Tokyo
  - Site Reference ID/Investigator# 41230, Tokyo
  - Site Reference ID/Investigator# 41239, Tokyo
  - Site Reference ID/Investigator# 41240, Tokyo
  - Site Reference ID/Investigator# 41241, Tokyo
  - Site Reference ID/Investigator# 41242, Tokyo
  - Site Reference ID/Investigator# 41243, Tokyo
  - Site Reference ID/Investigator# 41244, Tokyo
  - Site Reference ID/Investigator# 41245, Tokyo
  - Site Reference ID/Investigator# 41246, Tokyo
  - Site Reference ID/Investigator# 41259, Tokyo
  - Site Reference ID/Investigator# 41268, Tokyo
  - Site Reference ID/Investigator# 41273, Tokyo
  - Site Reference ID/Investigator# 41443, Tokyo
  - Site Reference ID/Investigator# 41444, Tokyo
  - Site Reference ID/Investigator# 41445, Tokyo
  - Site Reference ID/Investigator# 41446, Tokyo
  - Site Reference ID/Investigator# 41447, Tokyo
  - Site Reference ID/Investigator# 41448, Tokyo
  - Site Reference ID/Investigator# 41449, Tokyo
  - Site Reference ID/Investigator# 41459, Tokyo
  - Site Reference ID/Investigator# 41470, Tokyo
  - Site Reference ID/Investigator# 41474, Tokyo
  - Site Reference ID/Investigator# 41547, Tokyo
  - Site Reference ID/Investigator# 41602, Tokyo
  - Site Reference ID/Investigator# 41610, Tokyo
  - Site Reference ID/Investigator# 41742, Tokyo
  - Site Reference ID/Investigator# 41764, Tokyo
  - Site Reference ID/Investigator# 41765, Tokyo
  - Site Reference ID/Investigator# 41792, Tokyo
  - Site Reference ID/Investigator# 41795, Tokyo
  - Site Reference ID/Investigator# 41882, Tokyo
  - Site Reference ID/Investigator# 41883, Tokyo
  - Site Reference ID/Investigator# 41886, Tokyo
  - Site Reference ID/Investigator# 41887, Tokyo
  - Site Reference ID/Investigator# 41888, Tokyo
  - Site Reference ID/Investigator# 41890, Tokyo
  - Site Reference ID/Investigator# 41891, Tokyo
  - Site Reference ID/Investigator# 41892, Tokyo
  - Site Reference ID/Investigator# 41896, Tokyo
  - Site Reference ID/Investigator# 41897, Tokyo
  - Site Reference ID/Investigator# 41907, Tokyo
  - Site Reference ID/Investigator# 41911, Tokyo
  - Site Reference ID/Investigator# 41912, Tokyo
  - Site Reference ID/Investigator# 41913, Tokyo
  - Site Reference ID/Investigator# 41924, Tokyo
  - Site Reference ID/Investigator# 41925, Tokyo
  - Site Reference ID/Investigator# 56092, Tokyo
  - Site Reference ID/Investigator# 56093, Tokyo
  - Site Reference ID/Investigator# 56102, Tokyo
  - Site Reference ID/Investigator# 56104, Tokyo
  - Site Reference ID/Investigator# 56125, Tokyo
  - Site Reference ID/Investigator# 56126, Tokyo
  - Site Reference ID/Investigator# 56211, Tokyo
  - Site Reference ID/Investigator# 56225, Tokyo
  - Site Reference ID/Investigator# 56243, Tokyo
  - Site Reference ID/Investigator# 56244, Tokyo
  - Site Reference ID/Investigator# 56245, Tokyo
  - Site Reference ID/Investigator# 56246, Tokyo
  - Site Reference ID/Investigator# 56247, Tokyo
  - Site Reference ID/Investigator# 56248, Tokyo
  - Site Reference ID/Investigator# 56331, Tokyo
  - Site Reference ID/Investigator# 60000, Tokyo
  - Site Reference ID/Investigator# 60002, Tokyo
  - Site Reference ID/Investigator# 60008, Tokyo
  - Site Reference ID/Investigator# 60020, Tokyo
  - Site Reference ID/Investigator# 80885, Tokyo
  - Site Reference ID/Investigator# 80888, Tokyo
  - Site Reference ID/Investigator# 41787, Tonami
  - Site Reference ID/Investigator# 67142, Toride
  - Site Reference ID/Investigator# 56262, Tottori
  - Site Reference ID/Investigator# 41325, Toyama
  - Site Reference ID/Investigator# 41609, Toyama
  - Site Reference ID/Investigator# 41685, Toyama
  - Site Reference ID/Investigator# 41688, Toyama
  - Site Reference ID/Investigator# 41692, Toyama
  - Site Reference ID/Investigator# 41783, Toyama
  - Site Reference ID/Investigator# 56097, Toyama
  - Site Reference ID/Investigator# 56192, Toyama
  - Site Reference ID/Investigator# 56258, Toyama
  - Site Reference ID/Investigator# 60004, Toyama
  - Site Reference ID/Investigator# 64806, Toyama
  - Site Reference ID/Investigator# 41288, Toyoake
  - Site Reference ID/Investigator# 60010, Toyoake
  - Site Reference ID/Investigator# 67147, Toyoake
  - Site Reference ID/Investigator# 41307, Toyohashi
  - Site Reference ID/Investigator# 41845, Toyooka
  - Site Reference ID/Investigator# 56228, Toyooka
  - Site Reference ID/Investigator# 56089, Toyota
  - Site Reference ID/Investigator# 56114, Tsukuba
  - Site Reference ID/Investigator# 56115, Tsukuba
  - Site Reference ID/Investigator# 56204, Tsuyama
  - Site Reference ID/Investigator# 56210, Uji
  - Site Reference ID/Investigator# 41453, Urayasu
  - Site Reference ID/Investigator# 41759, Urayasu
  - Site Reference ID/Investigator# 41807, Utazu
  - Site Reference ID/Investigator# 41923, Utazu
  - Site Reference ID/Investigator# 80913, Utsunomiya
  - Site Reference ID/Investigator# 41463, Wakayama
  - Site Reference ID/Investigator# 41677, Wakayama
  - Site Reference ID/Investigator# 41681, Wakayama
  - Site Reference ID/Investigator# 41770, Wakayama
  - Site Reference ID/Investigator# 80890, Yachiyo
  - Site Reference ID/Investigator# 80891, Yachiyo
  - Site Reference ID/Investigator# 80894, Yachiyo
  - Site Reference ID/Investigator# 41894, Yamagata
  - Site Reference ID/Investigator# 41895, Yamagata
  - Site Reference ID/Investigator# 41898, Yamagata
  - Site Reference ID/Investigator# 56110, Yamagata
  - Site Reference ID/Investigator# 56328, Yamagata
  - Site Reference ID/Investigator# 41711, Yamaguchi
  - Site Reference ID/Investigator# 41722, Yamaguchi
  - Site Reference ID/Investigator# 41726, Yamaguchi
  - Site Reference ID/Investigator# 56199, Yamaguchi
  - Site Reference ID/Investigator# 56223, Yamaguchi
  - Site Reference ID/Investigator# 41899, Yamanashi
  - Site Reference ID/Investigator# 41297, Yatomi
  - Site Reference ID/Investigator# 41275, Yokohama
  - Site Reference ID/Investigator# 41276, Yokohama
  - Site Reference ID/Investigator# 41277, Yokohama
  - Site Reference ID/Investigator# 41285, Yokohama
  - Site Reference ID/Investigator# 41286, Yokohama
  - Site Reference ID/Investigator# 41450, Yokohama
  - Site Reference ID/Investigator# 41860, Yokohama
  - Site Reference ID/Investigator# 41916, Yokohama
  - Site Reference ID/Investigator# 56128, Yokohama
  - Site Reference ID/Investigator# 56332, Yokohama
  - Site Reference ID/Investigator# 71459, Yokohama
  - Site Reference ID/Investigator# 80917, Yokohama
  - Site Reference ID/Investigator# 41291, Yokosuka
  - Site Reference ID/Investigator# 71458, Yokosuka
  - Site Reference ID/Investigator# 41706, Yonago
  - Site Reference ID/Investigator# 41738, Yufu

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-four participants entered this study from study NCT00647400 (M04-702), a Phase III extension study of Humira (adalimumab) in Japan.
Pre-assignment Details: Of the 752 participants registered, 4 participants did not have case report forms retrieved (2 whose registration was duplicated and 2 who did not receive Humira). Of the remaining 748 participants, 14 were excluded from analysis (7 changed hospital after registration, 7 didn't visit clinic after the first Humira administration).
Period: Overall Study
Arm/Group | Humira
Started | 734 (Safety Analysis Population)
Efficacy Analysis Population | 708 (5 received Humira off-label, 21 did not receive Humira after the first administration)
Completed | 592
Not Completed | 142
Not completed — Adverse Event | 39
Not completed — Lack of Efficacy | 46
Not completed — Participant's Economic Reasons | 17
Not completed — No Hospital Visits | 7
Not completed — Adverse Event + Lack of Efficacy | 2
Not completed — Adverse Event + Other Reasons | 7
Not completed — Participant's Economic Reasons + Other | 1
Not completed — Other Reasons | 23

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population
Arm/Group | Humira
Number analyzed (Participants) | 734
Age Continuous [Mean (Standard Deviation); unit: years] | 50.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176
  Male | 558
Physician's Global Assessment (PGA) [Mean (Standard Deviation); unit: units on a scale] — The Physician's Global Assessment (PGA) is a 6-point scale used to measure the severity of disease at the time of the physician's evaluation of the participant. The degree of overall lesion severity was evaluated using the following categories: 0 (Clear); 1 (Minimal); 2 (Mild); 3 (Moderate); 4 (Severe); 5 (Very Severe). PGA was assessed at baseline in 644 participants.
  units on a scale | 2.7 (5.7)
Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions, and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI was assessed at baseline in 625 participants.
  units on a scale | 15.7 (12.2)
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: units on a scale] — Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each question are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. DLQI was assessed at baseline in 280 participants.
  units on a scale | 8.43 (6.77)
Pain Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — Participants assessed their pain due to psoriatic arthritis in the last week, on a a single-line Visual Analogue Scale (VAS) from 0 (no pain) to 100 (pain as bad as it could be). VAS was assessed at baseline in 153 participants.
  units on a scale | 49.5 (30.7)
Disease Activity Score 28-4, Erythrocyte Sedimentation Rate (DAS28-4 [ESR]) [Mean (Standard Deviation); unit: units on a scale] — DAS28-4 (ESR) is calculated using the number of tender and swollen joints (out of 28 counted), erythrocyte sedimentation rate (ESR), and the patient's global assessment of disease activity via the visual analog scale (VAS). The calculated range of DAS28-4 is 0.49 to 9.07. A DAS28-4 score less than 2.6 indicates clinical remission, DAS28-4 2.6 to 3.2 indicates low disease activity, DAS28-4 3.2 to less than 5.1 indicates moderate disease activity, and DAS28-4 of 5.1 or greater indicates high disease activity. DAS28-4 (ESR) was assessed at baseline in 94 participants with psoriatic arthritis.
  units on a scale | 4.4 (1.7)
Disease Activity Score 28-4, C-reactive Protein (DAS28-4 [CRP]) [Mean (Standard Deviation); unit: units on a scale] — DAS28-4 (CRP) is calculated using the number of tender and swollen joints (out of 28 counted), C-reactive protein (CRP) level, and the patient's global assessment of disease activity via the visual analog scale (VAS). The calculated range of DAS28-4 is 0.49 to 9.07. A DAS28-4 score less than 2.6 indicates clinical remission, DAS28-4 2.6 to 3.2 indicates low disease activity, DAS28-4 3.2 to less than 5.1 indicates moderate disease activity, and DAS28-4 of 5.1 or greater indicates high disease activity. DAS28-4 (CRP) was assessed at baseline in 131 participants with psoriatic arthritis.
  units on a scale | 3.5 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Drug Reactions (ADRs), Serious Adverse Drug Reactions (SADRs), Deaths, and Discontinuations Due to AEs
Description: This study was mandated by the Japanese government as an approval condition for Humira in Japan; therefore, definitions of adverse events and seriousness criteria were applicable as specified in the Japanese local standard operating procedures, based on local Japanese regulations. ADRs were defined as adverse events for which the causal relationship with Humira was other than "not related" (ie, "probable," "possible," or "unclear"). The count of participants with AEs presented in this table includes serious and nonserious AEs. The count of participants with discontinuations due to AEs includes those who discontinued due to an AE plus other reasons. Please see Safety section for further details regarding adverse events.
Time Frame: From study registration through Week 24
Population: Safety Analysis Population
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 734
participants
  AEs | 237
  SAEs | 35
  ADRs | 191
  SADRs | 24
  Deaths | 4
  Discontinuations Due to AEs | 48

2. Primary Outcome: Physician's Global Assessment at Week 4
Description: The Physician's Global Assessment (PGA) is a 6-point scale used to measure the severity of disease at the time of the physician's evaluation of the participant. The degree of overall lesion severity was evaluated using the following categories:
  * 0 / Clear (plaque elevation=none, scaling=none, erythema=hyperpigmentation, pigmented macules, diffuse faint pink or red coloration);
  * 1 / Minimal (plaque elevation=possible but difficult to ascertain whether there is a slight elevation above normal skin, scaling=surface dryness with some white coloration, erythema=up to moderate);
  * 2 / Mild (plaque elevation=slight, scaling=fine, erythema=up to moderate);
  * 3 / Moderate (plaque elevation=moderate, scaling=coarser, erythema=moderate);
  * 4 / Severe (plaque elevation=marked, scaling=coarse, erythema=severe);
  * 5 / Very Severe (plaque elevation=very marked, scaling=very coarse, erythema=very severe).
Time Frame: Week 4
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 640
units on a scale | 2.2 (1.1)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 4; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Primary Outcome: Physician's Global Assessment At Week 8
Description: as for outcome 2
Time Frame: Week 8
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 591
units on a scale | 1.8 (1.1)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 8; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Primary Outcome: Physician's Global Assessment at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 550
units on a scale | 1.5 (1.1)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 16; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

5. Primary Outcome: Physician's Global Assessment at Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 502
units on a scale | 1.2 (1.1)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Primary Outcome: Psoriasis Area and Severity Index (PASI) at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
Time Frame: Week 16
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 522
units on a scale | 5.0 (7.3)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 16; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

7. Primary Outcome: Psoriasis Area and Severity Index (PASI) at Week 24
Description: as for outcome 6
Time Frame: Week 24
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 476
units on a scale | 4.0 (7.4)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

8. Primary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 75 (PASI75) Response at Week 16
Description: PASI75 is defined as at least a 75% reduction in PASI (Psoriasis Area and Severity Index) score compared with the Baseline PASI score. PASI scores range from 0 (best) to 72 (worst), with the highest score representing complete erythroderma of the severest degree. The percent decrease in score is calculated as (Week 0 PASI score minus Week 16 PASI score) divided by Week 0 PASI score.
Time Frame: Baseline and Week 16
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Number; unit: percentage of participants
Groups:
- Humira (All Participants): Humira 40 mg (marketed product) every other week (eow) for subcutaneous injection after initial dosage of 80 mg.
- Humira (Adalimumab-naive Participants): Humira 40 mg (marketed product) every other week (eow) for subcutaneous injection after initial dosage of 80 mg. Excludes participants previously enrolled in study NCT00647400 (M04-072).
Arm/Group | Humira (All Participants) | Humira (Adalimumab-naive Participants)
Number analyzed (Participants) | 522 | 463
percentage of participants | 49.2 | 52.9

9. Primary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 75 (PASI75) Response at Week 24
Description: PASI75 is defined as at least a 75% reduction in PASI (Psoriasis Area and Severity Index) score compared with the Baseline PASI score. PASI scores range from 0 (best) to 72 (worst), with the highest score representing complete erythroderma of the severest degree. The percent decrease in score is calculated as (Week 0 PASI score minus Week 24 PASI score) divided by Week 0 PASI score.
Time Frame: Baseline and Week 24
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Number; unit: percentage of participants
Arm/Group | Humira (All Participants) | Humira (Adalimumab-naive Participants)
Number analyzed (Participants) | 476 | 422
percentage of participants | 58.2 | 62.1

10. Primary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 90 (PASI90) Response at Week 16
Description: PASI90 is defined as at least a 90% reduction in PASI (Psoriasis Area and Severity Index) score compared with the Baseline PASI score. PASI scores range from 0 (best) to 72 (worst), with the highest score representing complete erythroderma of the severest degree. The percent decrease in score is calculated as (Week 0 PASI score minus Week 16 PASI score) divided by Week 0 PASI score.
Time Frame: Baseline and Week 16
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Number; unit: percentage of participants
Arm/Group | Humira (All Participants) | Humira (Adalimumab-naive Participants)
Number analyzed (Participants) | 522 | 463
percentage of participants | 27.0 | 28.7

11. Primary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 90 (PASI90) Response at Week 24
Description: PASI90 is defined as at least a 90% reduction in PASI (Psoriasis Area and Severity Index) score compared with the Baseline PASI score. PASI scores range from 0 (best) to 72 (worst), with the highest score representing complete erythroderma of the severest degree. The percent decrease in score is calculated as (Week 0 PASI score minus Week 24 PASI score) divided by Week 0 PASI score.
Time Frame: Baseline and Week 24
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Number; unit: percentage of participants
Arm/Group | Humira (All Participants) | Humira (Adalimumab-naive Participants)
Number analyzed (Participants) | 476 | 422
percentage of participants | 39.3 | 41.7

12. Primary Outcome: Dermatology Life Quality Index at Week 16
Description: Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot (score of 2), a little (score of 1), or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired.
Time Frame: Week 16
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 205
units on a scale | 3.01 (4.51)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 16; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

13. Primary Outcome: Dermatology Life Quality Index at Week 24
Description: as for outcome 12
Time Frame: Week 24
Population: Observed cases: participants in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 193
units on a scale | 2.30 (3.89)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

14. Primary Outcome: Pain Visual Analog Scale (VAS) at Week 4
Description: Participants assessed their pain due to psoriatic arthritis in the past week, on a single-line Visual Analog Scale (VAS) from 0 (no pain) to 100 (pain as bad as it could be).
Time Frame: Week 4
Population: Observed cases: participants with psoriatic arthritis in the Efficacy Analysis Population with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 133
units on a scale | 26.7 (26.3)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 4; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

15. Primary Outcome: Pain Visual Analog Scale (VAS) at Week 16
Description: as for outcome 14
Time Frame: Week 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 111
units on a scale | 21.3 (23.7)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 16; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

16. Secondary Outcome: Physician's Overall Response Rating At Week 24
Description: Overall response rating, according to investigator's subjective clinical opinion. The level of overall improvement rating was categorized as "markedly improved," "improved," "not changed," or "not assessable," comparing clinical conditions at Week 24 or at discontinuation with Baseline conditions.
Time Frame: Baseline and Week 24
Population: Participants in the Efficacy Analysis Population with assessment at Week 24.
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 700
participants
  Markedly improved | 354
  Improved | 255
  Not changed | 65
  Aggravated | 16
  Not assessable | 10

17. Primary Outcome: Pain Visual Analog Scale (VAS) at Week 24
Description: as for outcome 14
Time Frame: Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 116
units on a scale | 16.3 (21.3)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

18. Primary Outcome: Disease Activity Score 28-4, Erythrocyte Sedimentation Rate (DAS28-4 [ESR]) at Week 4
Description: DAS28-4 (ESR) is calculated using the number of tender and swollen joints (out of 28 counted), erythrocyte sedimentation rate (ESR), and the patient's global assessment of disease activity via the visual analog scale (VAS). The calculated range of DAS28-4 is 0 to 10. A score less than 2.6 indicates clinical remission, a score of 2.6 to 3.2 indicates low disease activity, a score of 3.2 to less than 5.1 indicates moderate disease activity, and a score of 5.1 or greater indicates high disease activity.
Time Frame: Week 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 69
units on a scale | 3.0 (1.6)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 4; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

19. Primary Outcome: Disease Activity Score 28-4, Erythrocyte Sedimentation Rate (DAS28-4 [ESR]) at Week 16
Description: as for outcome 18
Time Frame: Week 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 61
units on a scale | 2.4 (1.3)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 16; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

20. Primary Outcome: Disease Activity Score 28-4, Erythrocyte Sedimentation Rate (DAS28-4 [ESR]) at Week 24
Description: as for outcome 18
Time Frame: Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 62
units on a scale | 2.3 (1.3)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

21. Primary Outcome: Disease Activity Score 28-4, C-reactive Protein (DAS28-4 [CRP]) at Week 4
Description: DAS28-4 (CRP) is calculated using the number of tender and swollen joints (out of 28 counted), C-reactive protein (CRP) level, and the patient's global assessment of disease activity via the visual analog scale (VAS). The calculated range of DAS28-4 is 0 to 10. A score less than 2.6 indicates clinical remission, a score of 2.6 to 3.2 indicates low disease activity, a score of 3.2 to less than 5.1 indicates moderate disease activity, and a score of 5.1 or greater indicates high disease activity.
Time Frame: Week 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 97
units on a scale | 2.3 (1.2)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 4; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

22. Primary Outcome: Disease Activity Score 28-4, C-reactive Protein (DAS28-4 [CRP]) at Week 16
Description: as for outcome 21
Time Frame: Week 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 82
units on a scale | 2.0 (0.9)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 16; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

23. Primary Outcome: Disease Activity Score 28-4, C-reactive Protein (DAS28-4 [CRP]) at Week 24
Description: as for outcome 21
Time Frame: Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 85
units on a scale | 1.8 (0.9)
Statistical Analysis 1: Comparison: Humira; comparison versus Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From study registration through Week 24
Description: Safety Analysis Population
Arm/Group | Humira
Serious Adverse Events (participants affected / at risk) | 35/734
Other Adverse Events (participants affected / at risk) | 0/734
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=734)
Diverticulitis (Infections and infestations) | 1
Encephalitis herpes (Infections and infestations) | 1
External ear cellulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Meningitis bacterial (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Esophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Cerebral hemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Temporal arteritis (Vascular disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Bleeding gastric ulcer (Gastrointestinal disorders) | 1
Pancreatic cyst (Gastrointestinal disorders) | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 3
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Chest pain (General disorders) | 1
Malaise (General disorders) | 1
Edema (General disorders) | 1
Pyrexia (General disorders) | 2
C-reactive protein increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.